CLINICAL TRIAL: NCT04399837
Title: Effisayil™ 2: Multi-center, Randomized, Parallel Group, Double Blind, Placebo Controlled, Phase IIb Dose-finding Study to Evaluate Efficacy and Safety of BI 655130 (Spesolimab) Compared to Placebo in Preventing Generalized Pustular Psoriasis (GPP) Flares in Patients With History of GPP.
Brief Title: A Study to Test Whether BI 655130 (Spesolimab) Prevents Flare-ups in Patients With Generalized Pustular Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0027; 2018-003081-14 (EudraCT Number)
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Spesolimab SC low dose (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab SC medium dose (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab SC high dose (Experimental)
  Interventions: Drug: Spesolimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab — Solution for injection
  Arms: Spesolimab SC high dose; Spesolimab SC low dose; Spesolimab SC medium dose
Drug: Placebo — Solution for injection
  Arms: Placebo

SUMMARY:
This is a study in adolescents and adults with Generalized Pustular Psoriasis (GPP). People between 12 and 75 years old can take part in the study. The study is open to people who had GPP flare-ups in the past but whose skin is clear or almost clear when they join the study. The purpose of the study is to test 3 different doses of a medicine called spesolimab and to see whether it helps to prevent GPP flare-ups.

Participants are put into 4 groups by chance. Three groups get different doses of spesolimab. The fourth group gets a placebo. Placebo looks like spesolimab but does not contain any medicine.

Spesolimab and placebo are given as an injection under the skin. Participants are in the study for about 1 year and 4 months. During this time, they visit the study site about 15 times. For the first 11 months, participants get spesolimab or placebo injections every month. At the study visits, the doctors check participants' skin for signs of a new GPP flare-up. The doctors also check the general health of the participants.

If a participant has a GPP flare-up during the study, more visits may be necessary. In case of a flare-up, participants get a dose of spesolimab as an infusion into a vein.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known and documented history of GPP per ERASPEN criteria (see Section 3.3.1) regardless of IL36RN mutation status, with at least 2 presentations of moderate to severe GPP flares with fresh pustulation (new appearance or worsening) in the past.
* Patients with a GPPGA score of 0 or 1 at screening and randomization.
* Patients who are not on concomitant GPP treatment at time of randomization (V2) must have had at least two presentations of moderate to severe GPP flare in the past year, at least one of which had evidence of either fever and/or elevated CRP and/or elevated WBC, and/or asthenia and/or myalgia.
* Patients who are not on concomitant GPP treatment at time of randomization (V2) but who were on concomitant GPP treatment until shortly before randomization (V2) (≤ 12 weeks before randomization), these patients must have a history of flaring while on concomitant treatment for GPP or in case of dose reduction or discontinuation of their concomitant medication.
* Patients who are on concomitant treatment regimen with retinoids and/or methotrexate and/or cyclosporine must stop at the day of randomization (V2). These patients must have a history of flaring while on concomitant treatment for GPP or in case of dose reduction or discontinuation of these concomitant medications.
* Male or female patients, aged 12 to 75 years at screening. For all patients, a minimum weight of 40 kg is required.
* Signed and dated written informed consent and assent in accordance with ICH-GCP and local legislation prior to admission in the trial.
* Women of childbearing potential (WOCBP)1 must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the CTP as well as in the patient, parent(s) (or patient's legal guardian) information.

Exclusion Criteria:

1. Patients with SAPHO (Synovitis-acne-pustulosis-hyperostosis-osteitis) syndrome.
2. Patients with primary erythrodermic psoriasis vulgaris.
3. Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold Upper Limit of Normal (ULN) elevation in Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin.
4. Treatment with:

   1. Any restricted medication as specified in the CTP, or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator.
   2. Any prior exposure to BI 655130 or another IL36R inhibitor biologic.
5. Increased risk of infectious complications (e.g. recent pyogenic infection, any congenital or acquired immunodeficiency (e.g. HIV), past organ or stem cell transplantation), as assessed by the investigator.
6. Relevant chronic or acute infections including active tuberculosis, human immunodeficiency virus (HIV) infection or viral hepatitis at the time of randomization. A patient can be re-screened if the patient was treated and is cured from the acute infection.
7. Active or Latent Tuberculosis (TB):

   * Patients with active tuberculosis should be excluded
   * Patients with a positive QuantiFERON® (or if applicable, T-Spot®) TB test during screening are excluded, unless the patient had previous diagnosis of active or latent TB and has completed appropriate treatment per the discretion of the local investigator within the last 3 years and at the latest at the time of screening (i.e. 2 to 4 weeks before study drug administration); patients may be re-screened once to meet this criterion)
   * Patients with suspected false positive or indeterminate QuantiFERON® (or if applicable, T-Spot®) TB result may be re-tested once
   * If QuantiFERON® (or if applicable, T-Spot®) TB testing is not available or provides indeterminate results after repeat testing, a tuberculin skin test (TST) can be performed: A TST reaction of ≥10mm (≥5mm if receiving ≥15mg/d prednisone or its equivalent) is considered positive.
8. History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients.

Further exclusion criteria apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (2):
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Washington University School of Medicine, St Louis, Missouri
- Argentina (2):
  - Buenos Aires Skin S.A., CABA
  - Hospital Italiano de Buenos Aires, CABA
- Brussels - UNIV Saint-Luc, Brussels, Belgium
- Clínica Dermacross S.A., Vitacura, Chile
- China (7):
  - Sun yet-sen Memorial Hospital, Sun yet-sen Univesity, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Shanghai Skin Disease Hospital, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
- France (2):
  - HOP l'Archet, Nice
  - HOP Saint-Louis, Paris
- Germany (7):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum der Universität München - Campus Innenstadt, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg AöR, Oldenburg
  - Universitätsklinikum Würzburg AÖR, Würzburg
- General Hospital of Thessaloniki "Ippokrateio", Thessaloniki, Greece
- Istituto Clinico Humanitas, Rozzano (MI), Italy
- Japan (6):
  - Nagoya City University Hospital, Aichi, Nagoya
  - Kyushu Rosai Hospital, Fukuoka, Kitakyushu
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki, Inashiki-gun
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
- Malaysia (8):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Sultan Ismail, Johor Bahru
  - Queen Elizabeth Hospital, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Pulau Pinang, Pulau Pinang
- Mexico (2):
  - Centro de Investigación de Enfermedades Autoinmunes S.C., Guadalajara
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Philippines (3):
  - Southern Philippines Medical Center, Davao City
  - Iloilo Doctors Hospital, Iloilo City, Iloilo
  - Center for Skin Research, Testing and Product Development, Makati City
- Russia (7):
  - SBHI Chelyabinsk Reg.Clin.Derma.Dispen., Chelyabinsk
  - LLC "Medical Center Azbuka Zdorovia", Kazan'
  - FSBEI HE "Kirov State Medical University", Kirov
  - LLC Skin Disease Clinic of Pier Volkenstein, St. Petersburg, Saint Petersburg
  - LLC "Avrora Medfort", Saint Petersburg
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - Saratov State Med.Univ.n.a.Razumovskogo, Saratov
- Arthritis Clinical Research Trials, Cape Town, South Africa
- South Korea (2):
  - Pusan National Univ. Hosp, Busan
  - Severance Hospital, Seoul
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues Del Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - Chang Gung Medical Foundation (CGMF) - Linkou Bran, Linkou District
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Institute of Dermatology, Bangkok
  - Ramathibodi Hospital, Ratchatewi, Bangkok
- Tunisia (5):
  - Hedi Chaker Hospital, Department of Dermatology, Sfax
  - Farhat Hached Hospital, Sousse
  - La Rabta Hospital, Tunis
  - Charles Nicolle Hospital, Tunis
  - Habib Thameur Hospital, Tunis
- Turkey (Türkiye) (4):
  - Uludag University Medicine Faculty Departmant of Dermatology, Bursa
  - Bezmi Alem Valide Sultan Vakif Gureba Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Marmara Universitesi Tip Fakultesi, Istanbul
- Vietnam (2):
  - National Hospital of Dermatology and Venereology, Hà Nội
  - HCMC Hospital of Dermato-Venereology, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Morita A, Choon SE, Bachelez H, Anadkat MJ, Marrakchi S, Zheng M, Tsai TF, Turki H, Hua H, Rajeswari S, Thoma C, Burden AD. Design of Effisayil 2: A Randomized, Double-Blind, Placebo-Controlled Study of Spesolimab in Preventing Flares in Patients with Generalized Pustular Psoriasis. Dermatol Ther (Heidelb). 2023 Jan;13(1):347-359. doi: 10.1007/s13555-022-00835-6. Epub 2022 Nov 5. PMID 36333618
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized multicenter, parallel group, double-blind, placebo-controlled Phase IIb trial comprising of 3 active doses compared to placebo in adolescents from 12 years to less than 18 years of age and adult patients with history of Generalized Pustular Psoriasis (GPP) and presenting (at screening and at randomization) with a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) score of 0 or 1 (clear or almost clear).
Pre-assignment Details: Subjects were screened for eligibility prior to participation and attended a specialist site which ensured that they (the subjects) met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
  The randomization was stratified accounting for use of systemic GPP medications at randomization (yes vs. no), and the blocking factors, region (Japan vs. non-Japan) and population (adults vs. adolescents).
Groups:
- Placebo: Patients were subcutaneously (SC) injected on Day 1 of Week 1 a loading dose of solution for injection of placebo matching solution for injection of spesolimab followed by a maintenance treatment which consisted of a subcutaneous injection of solution for injection of placebo matching solution for injection of spesolimab every 4 weeks (i.e. on Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 and 44).
  The patients who experienced a flare during the 48 week randomised treatment period were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at Day 1 of flare (R1/D1) or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare followed by OL maintenance treatment if time allowed which consisted of 300 mg of spesolimab administered SC every 12 weeks or every 4 weeks (intensified maintenance therapy).
- Spesolimab SC Low Dose: Patients received on Day 1 of Week 1 a loading dose which consisted of two subcutaneous (SC) injections of 150 mg of solution for injection of spesolimab (total dose of spesolimab=300mg) and two subcutaneous injections of placebo matching solution for injection of spesolimab. The loading dose was followed by a maintenance treatment which consisted of one SC injection of 150 mg of solution for injection of spesolimab and one SC injection of placebo matching solution for injection of spesolimab every 12 weeks (i.e. at Week 12, 24 and 36). To maintain the treatment blind during the trial the patients in this arm received two SC injections of placebo matching solution for injection of spesolimab at Week 4, 8, 16, 20, 28, 32, 40 and 44. The patients who experienced a flare during the 48 week randomised treatment period were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at Day 1 (R1/D1) of flare or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare followed by OL maintenance treatment if time allowed which consisted of 300 mg of spesolimab administered SC every 12 weeks or every 4 weeks (intensified maintenance therapy).
- Spesolimab SC Medium Dose: Patients received on Day 1 of Week 1 a loading dose which consisted of four subcutaneous (SC) injections of 150 mg of solution for injection of spesolimab (total dose of spesolimab= 600 mg). The loading dose was followed by a maintenance treatment which consisted of two SC injections of 150 mg of solution for injection of spesolimab (total dose of spesolimab=300 mg) every 12 weeks (i.e. at Week 12, 24 and 36). To maintain the treatment blind during the trial the patients in this arm received two SC injections of placebo matching solution for injection of spesolimab at Week 4, 8, 16, 20, 28, 32, 40 and 44. The patients who experienced a flare during the 48 week randomised treatment period were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at Day 1 (R1/D1) of flare or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare followed by OL maintenance treatment if time allowed which consisted of 300 mg of spesolimab administered subcutaneously every 12 weeks or every 4 weeks (intensified maintenance therapy).
- Spesolimab SC High Dose: Patients received on Day 1 of Week 1 a loading dose which consisted of four subcutaneous (SC) injections of 150 mg of solution for injection of spesolimab (total dose of spesolimab= 600 mg). The loading dose was followed by a maintenance treatment which consisted of two SC injections of 150 mg of solution for injection of spesolimab (total dose of spesolimab=300 mg) every 4 weeks (i.e. at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44). The patients who experienced a flare during the 48 week randomised treatment period were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at Day 1 (R1/D1) of flare or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare followed by OL maintenance treatment if time allowed which consisted of 300 mg of spesolimab administered SC every 12 weeks or every 4 weeks (intensified maintenance therapy).
Period: Overall Study
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Started | 31 | 31 | 31 | 30
Completed (Completed trial) | 30 | 27 | 28 | 26
Not Completed | 1 | 4 | 3 | 4
Not completed — Other than listed | 0 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set: This patient set includes all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose | Total
Number analyzed (Participants) | 31 | 31 | 31 | 30 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (14.0) | 38.9 (16.5) | 42.9 (16.7) | 40.2 (16.4) | 40.4 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 20 | 18 | 76
  Male | 13 | 11 | 11 | 12 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 1 | 7
  Not Hispanic or Latino | 28 | 28 | 31 | 29 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 17 | 20 | 21 | 21 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 14 | 11 | 10 | 9 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Number of patients in the categories 0 or 1 of GPPGA score [Count of Participants; unit: Participants] — Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) relied on the clinical assessment of GPP patient's skin presentation. The total score is calculated by taking the mean of the three subscores: 1) erythema; 2) pustules and 3) scaling/crusting which were assessed using a scale score 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score:
  0 , if scores for all three subscores are 0,
  1. if 0 < mean < 1.5;
  2. if 1.5 ≤ mean < 2.5;
  3. if 2.5 ≤ mean < 3.5;
  4. if mean ≥ 3.5. Number of patients in the categories 0 or 1 of GPPGA score is reported.
  Participants
    0 | 4 | 2 | 8 | 3 | 17
    1 | 27 | 29 | 23 | 27 | 106
Number of patients in the categories 0 or 1 of GPPGA pustules subscore [Count of Participants; unit: Participants] — The Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) pustules subscore relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) pustules presentation. The investigator (or qualified site personnel) scored the pustules of all GPP lesions from 0 to 4 where:
  0 = clear;
  1. = almost clear;
  2. = mild;
  3. = moderate;
  4. = severe. Number of patients in the categories 0 or 1 of GPPGA pustules subscore is reported.
  Participants
    0 | 21 | 23 | 24 | 20 | 88
    1 | 10 | 8 | 7 | 10 | 35
Concomitant use of systemic GPP medication at randomization [Count of Participants; unit: Participants] — Number of patients in each category of concomitant use of systemic GPP medication at randomization (-28 days to randomization). The reported categories of concomitant use of systemic GPP medication at randomization are:
  Yes; No.
  Participants
    No | 9 | 6 | 8 | 8 | 31
    Yes | 22 | 25 | 23 | 22 | 92
Psoriasis Symptom Scale (PSS) total score at baseline [Mean (Standard Deviation); unit: score on a scale] — The PSS is a 4-item patient-reported outcome (PRO) instrument that was developed to assess the severity of 4 psoriasis symptoms in patients with moderate to severe psoriasis.
  The symptoms included are: pain, redness, itching, and burning. Current symptom severity is assessed using a 5-point scale ranging from 0 (none) to 4 (very severe). The symptom scores are added to an unweighted total score (range: 0 (no symptoms) to 16 (severe symptoms). Population: Randomized Set: This patient set includes all randomized patients.
  score on a scale | 3.6 (2.9) | 4.1 (3.8) | 3.9 (2.9) | 5.3 (3.8) | 4.2 (3.4)
DLQI total score at baseline [Mean (Standard Deviation); unit: score on a scale] — The Dermatology Quality of Life Index (DLQI) is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Response categories range from 0 (not relevant) to 3 (very much). Question 7 is a "yes"/ "no" question where "yes" is scored as 3. Total score is obtained by summing the scores of each question resulting in a range of 0 (no effect on patient's life) to 30 (extremely large effect on patient's life). Population: This patient set includes all randomized patients. Adolescents aged below 16 years were optional to the questionnaire, therefore two adolescent whose age was below 16 years were not asked to fill this questionnaire.
  score on a scale
    number analyzed (Participants) | 31 | 30 | 31 | 29 | 121
    (all) | 7.2 (5.6) | 7.6 (6.7) | 6.6 (5.6) | 11.1 (6.9) | 8.1 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Generalized Pustular Psoriasis (GPP) Flare
Description: A GPP flare was defined as increase in Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) score by ≥ 2 from baseline and the pustular component of GPPGA ≥ 2) up to week 48. Use of rescue medication, or investigator-prescribed Standard of Care (SoC) for GPP worsening, was considered to represent a GPP flare onset.
  GPPGA relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The GPPGA total score was calculated by taking the mean of the erythema subscore, pustules subscore and scaling/crusting subscore. The severity of each subscore was assessed using a 5 point scale score ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score is assigned as follows:
  * 0 , if scores for all three subscores are 0,
  * 1, if 0 < mean < 1.5,
  * 2, if 1.5 ≤ mean < 2.5,
  * 3, if 2.5 ≤ mean < 3.5,
  * 4, if mean ≥ 3.5.
Time Frame: GPPGA was regularly assessed at baseline (Week 1) and up to Week 48 (at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48). Patients could come to site for flare confirmation anytime as unscheduled visit. Visit window was ±7 days.
Population: Randomized Set (EM-PM): This patient set includes all randomized patients. EM: Primary estimand for randomised maintenance period, where any use of rescue medication with intravenous spesolimab, or investigator-prescribed SoC for GPP worsening is considered as GPP flare. PM: Primary method for censoring, which is made at the earliest date of End of Study (EoS), Day 351 if no intercurrent event.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Number analyzed (Participants) | 31 | 31 | 31 | 30
weeks | 37.3 [4.0 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab SC Low Dose vs Spesolimab SC Medium Dose vs Spesolimab SC High Dose; A flat vs. non-flat dose-response relationship across the 3 doses of spesolimab and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 4 different plausible dose-response patterns (linear, Emax 1, Emax 2 and exponential) while protecting the overall probability of type I error (one-sided alpha of 0.05); Test type: Other — The generalized MCP-Mod procedure for time to event endpoints is based on the log hazard ratio of the active doses vs. placebo obtained via a Cox regression model on the time to first GPP flare; p = 0.002, MCP-Mod linear model fit; Model assumption: Dose effect is linear with the increase of dose; Multiple contrast test = 3.041
Statistical Analysis 2: Comparison: Placebo vs Spesolimab SC Low Dose vs Spesolimab SC Medium Dose vs Spesolimab SC High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, MCP-Mod Emax2 model fit; Model assumption: 95% of the maximum effect is achieved at low dose; Multiple contrast test = 3.033
Statistical Analysis 3: Comparison: Placebo vs Spesolimab SC Low Dose vs Spesolimab SC Medium Dose vs Spesolimab SC High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, MCP-Mod Emax1 model fit; Model assumption: 70% of the maximum effect is achieved at low dose; Multiple contrast test = 3.088
Statistical Analysis 4: Comparison: Placebo vs Spesolimab SC Low Dose vs Spesolimab SC Medium Dose vs Spesolimab SC High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, MCP-Mod exponential model fit; Model assumption: 35% of the maximum effect is achieved at medium dose; Multiple contrast test = 2.977
Statistical Analysis 5: Comparison: Placebo vs Spesolimab SC Medium Dose; Test type: Superiority — Null hypothesis: Effect of spesolimab 300 mg every 12 weeks on prolonging the time to the first GPP flare up to week 48 ≤ Placebo; p = 0.0269, Log Rank — One-sided p-value was computed from the log-rank test stratified by use of systemic GPP medication at randomisation. Threshold for statistical significance: one-sided p-value ≤ 0.01875; Hazard Ratio (HR) = 0.468, 95% CI 2-sided [0.206 to 1.064] — Hazard ratio and its 95% Confidence Interval are from Cox regression model stratified by use of systemic GPP medication at randomisation
Statistical Analysis 6: Comparison: Placebo vs Spesolimab SC High Dose; Test type: Superiority — Null hypothesis: Effect of spesolimab 300 mg every 4 weeks on prolonging the time to the first GPP flare up to week 48 ≤ Placebo; p = 0.0005, Log Rank — One-sided p-value is computed from the log-rank test stratified by use of systemic GPP medication at randomisation. Threshold for statistical significance: One-sided p-value ≤0.0125; Hazard Ratio (HR) = 0.157, 95% CI 2-sided [0.046 to 0.541] — Hazard ratio and its 95% CI (confidence interval) are from Cox regression model stratified by use of systemic GPP medication at randomisation

2. Secondary Outcome: Key Secondary Endpoint: The Occurrence of at Least One Generalized Pustular Psoriasis (GPP) Flare up to Week 48
Description: Proportion of patients with at least one GPP flare up to Week 48 is reported. Proportions were rounded up to three decimal places.
  A GPP flare was defined as increase in Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) score by ≥ 2 from baseline and the pustular component of GPPGA ≥ 2. Any use of rescue medication, or investigator-prescribed SoC for GPP worsening, prior to week 48 was considered to represent the onset of a GPP flare.
  Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) relied on the clinical assessment of GPP patient's skin presentation. The total score is calculated by taking the mean of the three subscores: 1) erythema; 2) pustules and 3) scaling/crusting which were assessed using a scale score 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score:
  0 , if scores for all three subscores are 0,
  1. if 0 < mean < 1.5;
  2. if 1.5 ≤ mean < 2.5;
  3. if 2.5 ≤ mean < 3.5;
  4. if mean ≥ 3.5.
Time Frame: as for outcome 1
Population: Randomized Set (EM-MI): This patient set includes all randomized patients. EM:primary estimand for randomised maintenance period, where any use of rescue medication with intravenous spesolimab, or investigator - prescribed SoC for GPP worsening is considered as GPP flare. MI: multiple imputation method using sequential logistic regression method.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Number analyzed (Participants) | 31 | 31 | 31 | 30
proportion of patients | 0.516 [0.348 to 0.680] | 0.226 [0.114 to 0.398] | 0.297 [0.181 to 0.445] | 0.127 [0.050 to 0.289]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab SC High Dose; Test type: Superiority — Null hypothesis: The proportion of patients who do not experience a GPP flare up to week 48 on BI 655130 300 mg every 4 weeks ≤ Placebo; p = 0.0013, Cochran-Mantel-Haenszel — One-sided p-value was computed from the Cochran-Mantel-Haenszel test stratified by use of systemic GPP medication at randomisation. one-sided alpha= 0.00625; Risk Difference (RD) = -0.390, 95% CI 2-sided [-0.621 to -0.159] — Risk difference=Spesolimab high dose-Placebo

3. Secondary Outcome: Time to First Worsening of Psoriasis Symptom Scale (PSS) up to Week 48
Description: Worsening of Psoriasis Symptom Scale (PSS) was defined as a 4-point increase in total score from baseline. Intake of rescue medication, or investigator-prescribed SoC for GPP worsening, was considered as onset of a worsening.
  The PSS is a 4-item patient-reported outcome (PRO) instrument that was developed to assess the severity of 4 psoriasis symptoms in patients with moderate to severe psoriasis.
  The symptoms included are: pain, redness, itching, and burning. Current symptom severity is assessed using a 5-point scale ranging from 0 (none) to 4 (very severe). The symptom scores are added to an unweighted total score (range: 0 (no symptoms) to 16 (severe symptoms)).
Time Frame: PSS assessments were performed at: Baseline (Week 1) and up to Week 48 (at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48). Visit window was ±7 days.
Population: Randomized Set (EM-PM): This patient set includes all randomized patients. EM:primary estimand for randomised maintenance period, where any use of rescue medication with intravenous spesolimab, or investigator-prescribed SoC for GPP worsening is considered as GPP flare. PM: primary method for censoring, which is made at the earliest date of End of Study (EoS), Day 351 if no intercurrent event.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Number analyzed (Participants) | 31 | 31 | 31 | 30
weeks | 16.0 [4.0 to NA] — Insufficient number of participants with events. | NA [8.1 to NA] — Insufficient number of participants with events. | NA [8.7 to NA] — Insufficient number of participants with events. | NA [12.0 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab SC High Dose; Hazard ratio and its 95% CI (confidence interval) are from Cox regression model stratified by use of systemic GPP medication at randomisation; Test type: Superiority — Null hypothesis: Effect of BI 655130 300 mg every 4 weeks on prolonging the time to first worsening of PSS up to week 48 ≤ Placebo; p = 0.0134, Log Rank — One-sided p-value was computed from the log-rank test stratified by use of systemic GPP medication at randomisation. one-sided alpha= 0.00625; Hazard Ratio (HR) = 0.424, 95% CI 2-sided [0.197 to 0.914] — spesolimab high dose vs. Placebo

4. Secondary Outcome: Time to First Worsening of Dermatology Quality of Life Index (DLQI) up to Week 48
Description: Worsening of DLQI up to week 48 was defined as a 4-point increase in total score from baseline. Intake of rescue medication, or investigator-prescribed SoC for GPP worsening, was considered as onset of a worsening.
  The DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Response categories include "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3). Question 7 is a "yes"/ "no" question where "yes" is scored as 3. DLQI total score is calculated by summing the scores of each question resulting in a range of 0 (no effect on patient's life) to 30 (extremely large effect on patient's life).
Time Frame: DLQI assessments were performed at: Baseline (Week 1) and up to Week 48 (at Week 4, 8, 12, 24, 36 and 48). Visit window was ±7 days. Time window for Week 48 was from Week 46 to Week 50.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Number analyzed (Participants) | 31 | 31 | 31 | 30
weeks | 16.0 [4.0 to NA] — Insufficient number of participants with events. | 35.8 [8.1 to NA] — Insufficient number of participants with events. | 49.3 [8.7 to 49.3] | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab SC High Dose; Hazard ratio and its 95% CI (confidence interval) are from Cox regression model stratified by use of systemic GPP medication at randomisation. one-sided alpha= 0.00625; Test type: Superiority — Null hypothesis: Effect of BI 655130 300 mg every 4 weeks on prolonging the time to the first worsening of DLQI up to week 48 ≤ Placebo; p = 0.0010, Log Rank — One sided p-value was computed from the log-rank test stratified by use of systemic GPP medication at randomisation; Hazard Ratio (HR) = 0.259, 95% CI 2-sided [0.109 to 0.620] — spesolimab high dose vs. Placebo

5. Secondary Outcome: Sustained Remission
Description: Proportion of patients with sustained remission at all visits up to Week 48. Proportions were rounded up to three decimal places.
  Remission was defined as a patient with a GPPGA score of 0 or 1 (clear or almost clear) at all visits up to week 48, without intake of rescue medication, or investigator-prescribed SoC for GPP worsening.
  GPPGA relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The GPPGA total score was calculated by taking the mean of the erythema subscore, pustules subscore and scaling/crusting subscore. The severity of each subscore was assessed using a 5 point scale score ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score is assigned as follows:
  * 0 , if scores for all three subscores are 0,
  * 1, if 0 < mean < 1.5,
  * 2, if 1.5 ≤ mean < 2.5,
  * 3, if 2.5 ≤ mean < 3.5,
  * 4, if mean ≥ 3.5.
Time Frame: as for outcome 1
Population: Randomized Set (EM-MI): This patient set includes all randomized patients. EM:primary estimand for randomised maintenance period, where any use of rescue medication with intravenous spesolimab, or investigator-prescribed SoC for GPP worsening is considered as GPP flare. MI: multiple imputation method using sequential logistic regression method.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose
Number analyzed (Participants) | 31 | 31 | 31 | 30
proportion of patients | 0.290 [0.161 to 0.466] | 0.516 [0.348 to 0.680] | 0.452 [0.292 to 0.622] | 0.633 [0.471 to 0.770]

6. Secondary Outcome: The Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of patients with treatment emergent adverse events (TEAEs) is reported. Percentages were rounded up to one decimal places.
  Time Frame: Placebo, Spesolimab (Speso) SC low, medium, high: From randomized study treatment start until the first use of rescue medication with IV spesolimab or until last dose + 16 weeks, up to 62 weeks.
  Speso IV SD and Speso IV DD: From first use of rescue medication with IV spesolimab until OL maintenance spesolimab SC or until last dose of spesolimab IV + 16 weeks, up to 17 weeks.
  Speso OL SC: From the first dose of OL spesolimab SC treatment until last dose + 16 weeks, up to 62 weeks.
Time Frame: Up to 62 weeks (for detailed timeframe see description).
Population: Arms "Placebo, Speso SC Low, medium, high":Safety Set (SAF)-This patient set included all patients who were randomized and received at least one dose of study drug. One patient who was randomized to placebo arm but received active spesolimab dose is reported under the arm "Spesolimab SC low" instead of "Placebo".
  Arms "Speso IV SD, Speso IV SD": Safety Analysis set for flare rescue treatment period (SAF-FT).
  Arm "Speso OL SC": Safety Analysis set for OL maintenance treatment period (SAF-MT).
Measure: Number; unit: percentage of patients
Groups:
- Spesolimab IV SD: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who took a single dose (SD) of rescue treatment of 900 milligram (mg) of spesolimab administered intravenously (IV) at Day 1 of flare (R1/D1) because of a GPP flare during the 48-week treatment randomised period.
- Spesolimab IV DD: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who took two doses (DD) of rescue treatment of spesolimab each 900 milligram (mg) of spesolimab administered intravenously (IV) at Day 1 and at Day 8 of flare (R1/D1 and R3/D8) because of a GPP flare during the 48-week treatment randomised period.
- Spesolimab OL SC: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who experienced a flare during the 48-week randomised treatment period and were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at either Day 1 (R1/D1) of flare or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare and then followed by maintenance treatment which consisted of 300 mg of spesolimab administered SC every 12 weeks or every 4 weeks (intensified maintenance therapy).
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose | Spesolimab IV SD | Spesolimab IV DD | Spesolimab OL SC
Number analyzed (Participants) | 30 | 32 | 31 | 30 | 22 | 10 | 20
percentage of patients | 86.7 | 90.6 | 93.5 | 86.7 | 68.2 | 60.0 | 75.0

ADVERSE EVENTS:
Time Frame: Placebo, Spesolimab (Speso) SC low, medium, high: From randomized study treatment start until the first use of rescue medication with IV spesolimab or until last dose + 16 weeks, up to 62 weeks. Speso IV SD and Speso IV DD: From first use of rescue medication with IV spesolimab until OL maintenance spesolimab SC or until last IV dose + 16 weeks, up to 17 weeks. Speso OL SC: From the first dose of OL spesolimab SC treatment until last dose + 16 weeks, up to 62 weeks.
Description: Arms "Placebo, Speso SC Low, medium, high":Safety Set (SAF)-This patient set included all patients who were randomized and received at least one dose of study drug. One patient who was randomized to placebo arm but received active spesolimab dose is reported under the arm "Spesolimab SC low" instead of "Placebo".
  Arms "Speso IV SD, Speso IV SD": SAF-FT- Safety Analysis set for flare rescue treatment period.
  Arm "Speso OL SC": SAF-MT- Safety Analysis set for OL maintenance treatment period.
Groups:
- Spesolimab IV SD: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who took a single dose (SD) of rescue treatment of 900 milligram (mg) of spesolimab administered intravenously (IV) at Day 1 of flare (R1/D1) because of a GPP flare during the 48 week treatment randomised period.
- Spesolimab IV DD: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who took two doses (DD) of rescue treatment of spesolimab each 900 milligram (mg) of spesolimab administered intravenously (IV) at Day 1 and at Day 8 of flare (R1/D1 and R3/D8) because of a GPP flare during the 48 week treatment randomised period.
- Spesolimab OL SC: This arm includes the patients who were randomized at study start in the arms "Placebo" or "Spesolimab SC low dose" or "Spesolimab SC medium dose" or "Spesolimab SC high dose" who experienced a flare during the 48 week randomised treatment period and were administered intravenously (IV) in an open label (OL) fashion with 900 milligram (mg) of solution for infusion of spesolimab at either Day 1 (R1/D1) of flare or at Day 1 (R1/D1) and at Day 8 (R3/D8) of flare and then followed by maintenance treatment which consisted of 300 mg of spesolimab administered SC every 12 weeks or every 4 weeks (intensified maintenance therapy).
Arm/Group | Placebo | Spesolimab SC Low Dose | Spesolimab SC Medium Dose | Spesolimab SC High Dose | Spesolimab IV SD | Spesolimab IV DD | Spesolimab OL SC
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32 | 0/31 | 0/30 | 0/22 | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/30 | 5/32 | 1/31 | 3/30 | 1/22 | 4/10 | 1/20
Other Adverse Events (participants affected / at risk) | 24/30 | 25/32 | 23/31 | 20/30 | 12/22 | 3/10 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Spesolimab SC Low Dose (N=32) | Spesolimab SC Medium Dose (N=31) | Spesolimab SC High Dose (N=30) | Spesolimab IV SD (N=22) | Spesolimab IV DD (N=10) | Spesolimab OL SC (N=20)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Spesolimab SC Low Dose (N=32) | Spesolimab SC Medium Dose (N=31) | Spesolimab SC High Dose (N=30) | Spesolimab IV SD (N=22) | Spesolimab IV DD (N=10) | Spesolimab OL SC (N=20)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 4 | 4 | 5 | 0 | 0 | 2
Injection site induration (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Injection site pain (General disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 2
Injection site swelling (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 2 | 2 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 1 | 3 | 0 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 6 | 0 | 1 | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 4 | 2 | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 2 | 4 | 1 | 0 | 0 | 0 | 0
Blood trypsin increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Tryptase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 3 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 2 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 4 | 5 | 4 | 1 | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 16 | 9 | 9 | 2 | 5 | 0 | 4
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT04399837/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04399837/SAP_001.pdf